CLINICAL TRIAL: NCT06772207
Title: Cardiac Rehabilitation Needs Among Individuals With Atrial Fibrillation. A Protocol for a Danish Survey and Registry-based Study (PRIME-AF)
Brief Title: Cardiac Rehabilitation Needs Among Individuals With Atrial Fibrillation
Acronym: PRIME-AF
Status: Enrolling by invitation | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Matilde Elnegaard, PhD student, Odense University Hospital
Other Study IDs: PRIME-AF
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Cardiac rehabilitation; Needs; Secondary prevention; Primary care; Survey; Registry
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Respondents of electronic survey: Population with incident AF in Denmark in 2023-2024

SUMMARY:
The goal of this survey- and registry-based study is to learn about the cardiac rehabilitation needs of individuals with atrial fibrillation (AF). The main objectives of the study is to:

1. Investigate cardiac rehabilitation needs among eligible individuals with AF in a large AF population
2. Estimate how many needs referral to primary care programs, according to a needs assessment model.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in adults globally. It poses significant public health challenges and is associated with substantial morbidity and mortality. AF affects quality of life with an enlarged symptom burden. To improve life expectancy and quality of life, medical treatment along with risk factor management and cardiac rehabilitation is needed. In many countries, referral to cardiac rehabilitation remains low. Furthermore, no guidelines or evidence provides details on whom should be referred. Thus, we do not know how many individuals with AF presents with cardiac rehabilitation needs.

This study is a survey and registry-based study. Danish health registries are used to draw a population of individuals with incident AF in 2023-2024. Following the exclusion criteria, these will receive a survey covering the described outcomes which are used to investigate needs of rehabilitation. A statistical predicitive analysis will be performed to estimate how many needs referral to cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with recidence in Denmark, 18 years of age or above, with a CPR number (personal identification number) registered with a diagnosis of incident AF in 2022 or 2023 (ICD-10: DI480*).

Exclusion Criteria:

* Death.
* Name- and address protection.
* Exemtion from using digital post.
* Living in a nursing home.
* A diagnosis of dementia.
* Hospital admission or ambulant contacts due to mental illness within one year before diagnosis (except depression or anxiety).
* Individuals receiving palliative care or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry-based. The study population is drawn from Danish Health Registries and receive an online questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation related quality of life | At enrollment
  Atrial fibrillation related quality of life by ASTA HRQoL scale (The Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmia).
  The ASTA HRQoL scale has 13 items and describes the arrhythmia's influence on daily life situation with a seven items physical subscale (items 1-5, 10 and 12) and a six items mental subscale (items 6-9, 11 and 13). We will be using both the total and subscale scores as recommended.
  The response alternatives from 0 to 3: "No (0), Yes, to a certain extent (1), Yes, quite a lot (2), Yes, a lot (3)". Scoring for the ASTA HRQoL total scale ranges from 0 (best possible HRQoL) to highest 39 (worst possible HRQoL). Higher scores reflect a worse effect on HRQoL due to the heart rhythm disturbance. ASTA's physical subscale ranges from 0 to 21 and the mental subscale ranges from 0 to18.
Atrial fibrillation related symptom burden | At enrollment
  AF6 questionnaire. Patients chose a number on a Likert scale from 0 to 10, where 0 means no and 10 severe symptoms or difficulties. The scores of the six questions are added into a single global score. The recall period for the instrument is the most recent 7 days.

SECONDARY OUTCOMES:
General well-being | At enrollment
  WHO5. The WHO-5 is a five-item scale measuring well-being and life satisfaction within the past 2 weeks and the scale is operationalized using a 0-100 score, with higher values indicating a higher level of well-being and life satisfaction. Scores below 50 indicate poor well-being.
Anxiety | At enrollment
  ASS-2 has the purpose of screening for anxiety within the past 2 weeks. Higher score of ASS-2 indicates a higher symptom level of anxiety.
Depression | At enrollment
  MDI-2 has the purpose of screening for depression within the past 2 weeks. Higher score indicates a higher symptom level of depression.
Medicine adherence | At enrollment
  MARS-5 (Medication Adherence Report Scale). Items scored as 5 = never to 1 = always, i.e. high scores = high adherence. Scores are added together to form a scale score (range = 5 to 25). An adjusted mean score is calculated by dividing the scale mean by the number of items in the scale (range 1-5).
Risk factor status | At enrollment
  Obesity, physical inactivity, smoking and alcohol habits
Comorbidity | At enrollment
  Hypertension, diabetes, sleep apnoea, other cardiac diseases

OTHER OUTCOMES:
General health status | At enrollment
  EQ-5D-5L. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state; for instance, 21111 means slight problems in the mobility dimension and no problems in any of the other dimensions. The EQ VAS records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). The EQ VAS provides a quantitative measure of the patient's perception of their overall health.
Demographic data | At enrollment
  Age, gender, civil status, living situation, region of Denmark, educational level, occupational status, ethnicity, socio-economic classification and family disposable income.
Outcomes important for the overall assessment of cardiac rehabilitation needs | At enrollment
  Questions regarding family relations, health literacy (HLS-EU-Q12), management of heart disease, previous provided information of cardiac rehabilitation and motivation for these interventions forwardly.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Brandes, Professor, cardiologist, Study Chair — Department of Cardiology, Esbjerg and Grindsted Hospital - University Hospital of Southern Denmark, Esbjerg, Denmark.
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
Unless follow-up studies using the same study population is planned later on, data (IPD) will not be shared.

REFERENCES:
- [Derived] Elnegaard CM, Borregaard B, Risom SS, Tveskov C, Bech M, von Bornemann Hjelmborg J, Eilso J, Hedegaard AM, Stege Bojer A, Darkner S, Albertsen AE, Joensen AM, Brandes A, Zwisler AD. Cardiac rehabilitation in atrial fibrillation: a protocol for a Danish survey and registry-based study (PRIME-AF). BMJ Open. 2025 Dec 24;15(12):e107042. doi: 10.1136/bmjopen-2025-107042. PMID 41448694